CLINICAL TRIAL: NCT04137718
Title: Multicenter Observational Study for Clinicopathological Characteristics and Clinical Efficacy of Chinese Non-Small Cell Lung Cancer (NSCLC) Patients With Rare Driver Gene Mutation
Brief Title: Multicenter Observational Study of Chinese Non-Small Cell Lung Cancer (NSCLC) Patients With Rare Driver Gene Mutation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Chief Physician, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: LC-IRICA
Record Dates: First submitted 2019-10-14; First posted 2019-10-24 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Chinese; Non-Small Cell Lung Cancer
Keywords: Multicenter; Observational Study; NSCLC; Rare Driver Gene
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rare driver gene mutation-positive: Screen the enrolled patients according to the admission criteria. The detection of lung cancer Polymerase Chain Reaction (PCR) panel kit in the hospital requires the use of tissue samples and the results show a rare driver gene mutation positive.
  Interventions: Other: nonIntervention
- Rare driver gene mutation-negative: Screen the enrolled patients according to the admission criteria. The detection of lung cancer Polymerase Chain Reaction(PCR)panel kit in the hospital requires the use of tissue samples and the results show a rare driver gene mutation negative.
  Interventions: Other: nonIntervention

INTERVENTIONS:
Other: nonIntervention — nonIntervention

SUMMARY:
Title: Multicenter observational study for clinicopathological characteristics and clinical efficacy of Chinese Non-Small Cell Lung Cancer (NSCLC) patients With Rare Driver Gene Mutation.

Purpose: To observe the status of rare driver gene mutations in NSCLC patients and identify the subtypes of the mutations.

By comparing and analyzing the relationship between different subtypes, clinicopathological features and clinical efficacy, to find out the effects on anti-tumor therapy and disease survival.

And ultimately to promote the precise application of clinical specifications for new anti-tumor drugs.

Study type: Observational

DETAILED DESCRIPTION:
Inclusion criteria:

1. Female or male, 18 years of age or older；
2. Histologically or cytologically proven diagnosis of NSCLC；
3. Able to get tumor tissue gene testing results by lung cancer Polymerase Chain Reaction(PCR)panel kit carried out in hospital
4. Signed and dated informed consent.

Exclusion criteria:

1. Combine with other tumor type
2. The investigator judges the situation that may affect the clinical search process and results.

Estimated enrollment: 50000 participants.

Outcome measures:

Primary outcome measures：

1. The NSCLC rare driver gene mutation frequency and clinicopathological features in 50,000 patients in real world;
2. The relationship between rare driver gene subtypes and clinicopathological features (age, gender, smoking history, histological subtype, clinical stage, lymph node metastasis, local metastasis, distant metastasis, brain metastasis) in NSCLC patients.

Secondary outcome measures:

1. The relationship between rare driver gene mutation subtypes and disease survival or prognosis (Objective response rate (ORR), Progression-free survival (PFS), and Overall survival (OS)) in NSCLC patients.

Method of Research:

1. Pre- entry/screening period (V0)

   1. Screen the enrolled patients according to the admission criteria. The detection of lung cancer PCR panel kit in the hospital requires the use of tissue samples (including surgical tissue, biopsy tissue under interventional conditions, lymph node biopsy tissue, metastases' tissue, etc.);
   2. All enrolled samples should be tested Neurotrophic-Tropomyosin Receptor Kinase (NTRK) gene mutation (PCR);
   3. If a)+b) results show a rare driver gene mutation was detected, participants will be involved into the next step; if a)+b) test results were negative, then 500 cases were selected for next generation sequencing (NGS) detection in this population, and were involved into the next step;
2. Baseline period (V1)

   a. Do further classification of rare driver gene mutation positive samples by Sanger sequencing, and record the test results;
3. Follow-up period (V2)

   1. Record the disease therapeutic regimen and follow-up of the survival status of the enrolled patients;
   2. Once every 3 months (or according to clinical needs) up to 60 months or death;
   3. Collect information including follow-up treatment, disease status, and survival status, imaging examination results, laboratory examination results, etc. (see the Case Report Form (CRF) form for details);
   4. For those who need further molecular testing (such as primary drug resistance), multi-gene analysis using the next generation sequencing (NGS) method;
   5. Loss of follow-up: If the patient fails to return to the center for a follow-up visit, the center will make two attempts to contact by phone and keep the contact records. If the patient does not respond within 1 month after the second contact, the patient is considered to have lost the interview.

Materials and Methods:

Materials:

The specimen material must be human genomic DNA and total RNA extracted from tumor tissue samples. Before the extraction of DNA and RNA, it is very important to make sure that there is at least 20% tumor cells in the tumor tissue samples.

Methods:

Epidermal Growth Factor Receptor 20 exon insertion (EGFR exon 20-ins) mutation/Activin Receptor-like Kinase (ALK) fusion/ROS proto-oncogene 1 receptor tyrosine kinase (ROS1) fusion/Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS) mutation/Neuroblastoma RAS viral oncogene homolog (NRAS) mutation/B-Raf proto-oncogene, serine/threonine kinase (BRAF) mutation/Phosphatidylinositol-4,5-bisphosphate 3-kinase catalytic subunit alpha (PIK3CA) mutation/RET proto-oncogene (RET) fusion/Mesenchymal-Epithelial Transition factor (MET) 14 exon skipping/Erb-b2 Receptor Tyrosine Kinase 2 (ERBB2) mutation/ Neurotrophic-Tropomyosin Receptor Kinase (NTRK) fusion mutation were detected by Fluorogenic Quantitative Polymerase Chain Reaction in Chinese NSCLC.

1. DNA/RNA Extraction:

   The total RNA concentration for gene fusion detection is 10~100 ng/µL in Formalin-Fixed Paraffin-Embedded (FFPE) tissue or 2~30 ng/µL in Fresh tissue.

   The amount of extracted DNA for gene mutation detection is 1.5~3 ng/µL in FFPE tissue or 0.5~1 ng/µL in Fresh tissue.
2. RNA Reverse Transcription.
3. Detection of the Target Alterations in RNA and DNA:

   ALK, ROS1, RET, NTRK Gene fusion and MET 14 exon skipping mutation were detected in RNA.

   EGFR 20 exon-ins, KRAS, NRAS, BRAF, PIK3CA and ERBB2 mutation were detected in DNA.
4. Result Interpretation

ELIGIBILITY:
Inclusion Criteria:

1. Female or male, 18 years of age or older；
2. Histologically or cytologically proven diagnosis of NSCLC；
3. Able to get tumor tissue gene testing results by lung cancer PCR panel kit carried out in hospital；
4. Signed and dated informed consent。

Exclusion Criteria:

1. Combine with other tumor type
2. The investigator judges the situation that may affect the clinical search process and results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically or cytologically proven diagnosis of NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2022-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Driver gene mutation frequency of Chinese NSCLC patients | 2022
  Analyze the rare driver gene mutation frequency in NSCLC patients in the real world.
Clinicopathological characteristics of Chinese NSCLC patients With Rare Driver Gene Mutation | 2022
  Observe the clinicopathological features in NSCLC patients with rare gene mutation in the real world.
Relationship of Clinicopathological characteristics and Rare Driver Gene Mutation of Chinese NSCLC patients | 2022
  Analyze the relationship between rare driver gene subtypes and clinicopathological features in NSCLC patients.

SECONDARY OUTCOMES:
Objective response rate of Chinese NSCLC patients With Rare Driver Gene Mutation | 2024
  The relationship between rare driver gene mutation subtypes and objective response rate in NSCLC patients.
  Objective response rate(ORR): ORR = (number of subjects with complete response (CR) + partial response (PR)) / total number of subjects × 100%, 95% confidence interval(CI) was calculated using binomial distribution, and the calculation of objective response rate was based on the quadratic confirmed optimal efficacy evaluation.
Progression-free survival of Chinese NSCLC patients With Rare Driver Gene Mutation | 2024
  The relationship between rare driver gene mutation subtypes and progression-free survival in NSCLC patients.
  Progression-free survival (PFS): PFS refers to the time (month) between the date of randomization to the first demonstration of disease progression or death (whichever occurs first).
Overall survival of Chinese NSCLC patients With Rare Driver Gene Mutation | 2024
  The relationship between rare driver gene mutation subtypes and overall survival in NSCLC patients.
  Overall survival (OS): OS refers to the time of first use of the drug to the time of death. At the end of the study, if the subject is still alive, refer the known "date of last survival of the subject" as the date of censoring.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wen S, Dai L, Wang L, Wang W, Wu D, Wang K, He Z, Wang A, Chen H, Zhang P, Dong X, Dong YA, Wang K, Yao M, Wang M. Genomic Signature of Driver Genes Identified by Target Next-Generation Sequencing in Chinese Non-Small Cell Lung Cancer. Oncologist. 2019 Nov;24(11):e1070-e1081. doi: 10.1634/theoncologist.2018-0572. Epub 2019 Mar 22. PMID 30902917
- [Result] Yasuda H, Park E, Yun CH, Sng NJ, Lucena-Araujo AR, Yeo WL, Huberman MS, Cohen DW, Nakayama S, Ishioka K, Yamaguchi N, Hanna M, Oxnard GR, Lathan CS, Moran T, Sequist LV, Chaft JE, Riely GJ, Arcila ME, Soo RA, Meyerson M, Eck MJ, Kobayashi SS, Costa DB. Structural, biochemical, and clinical characterization of epidermal growth factor receptor (EGFR) exon 20 insertion mutations in lung cancer. Sci Transl Med. 2013 Dec 18;5(216):216ra177. doi: 10.1126/scitranslmed.3007205. PMID 24353160
- [Result] Du X, Shao Y, Qin HF, Tai YH, Gao HJ. ALK-rearrangement in non-small-cell lung cancer (NSCLC). Thorac Cancer. 2018 Apr;9(4):423-430. doi: 10.1111/1759-7714.12613. Epub 2018 Feb 28. PMID 29488330
- [Result] Lin JJ, Shaw AT. Recent Advances in Targeting ROS1 in Lung Cancer. J Thorac Oncol. 2017 Nov;12(11):1611-1625. doi: 10.1016/j.jtho.2017.08.002. Epub 2017 Aug 14. PMID 28818606
- [Result] Lee CK, Man J, Lord S, Cooper W, Links M, Gebski V, Herbst RS, Gralla RJ, Mok T, Yang JC. Clinical and Molecular Characteristics Associated With Survival Among Patients Treated With Checkpoint Inhibitors for Advanced Non-Small Cell Lung Carcinoma: A Systematic Review and Meta-analysis. JAMA Oncol. 2018 Feb 1;4(2):210-216. doi: 10.1001/jamaoncol.2017.4427. PMID 29270615
- [Result] Zhou F, Zhou C. Lung cancer in never smokers-the East Asian experience. Transl Lung Cancer Res. 2018 Aug;7(4):450-463. doi: 10.21037/tlcr.2018.05.14. PMID 30225210
- [Result] Drilon A, Hu ZI, Lai GGY, Tan DSW. Targeting RET-driven cancers: lessons from evolving preclinical and clinical landscapes. Nat Rev Clin Oncol. 2018 Mar;15(3):150. doi: 10.1038/nrclinonc.2017.188. Epub 2017 Nov 28. PMID 29182164